CLINICAL TRIAL: NCT00291408
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Effect of Symbicort® and Pulmicort® on HAT and HDAC Expression and Activity in Induced Sputum Cells Obtained From COPD Patients.
Brief Title: Effect of Symbicort on HAT and HDAC in Sputum Macrophages of COPD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Researchers left the institute
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 05/Q0403/171; EudraCT Number: 2005-003297-13
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Age Matched Healthy Volunteers (Non-smokers)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Patch Tests

INTERVENTIONS:
Procedure: Skin Prick Test
Procedure: Impulse Oscillometry
Procedure: Exhaled Nitric Oxide
Procedure: Spirometry
Procedure: Reversibility
Procedure: Exhaled Breath Condensate
Procedure: Sputum Induction

SUMMARY:
The purpose of the study is to compare histone acetyltransferase (HAT) and histone deacetylase (HDAC) expressions and activities in induced sputum macrophages obtained from patients with moderate to severe COPD and age-matched normal non-smokers

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria-Healthy non-smokers

* Non-smoking volunteer
* aged 40 -75 years (age matched to COPD patients)
* Normal spirometry (normal FEV1/FVC ratio >70% and FEV1>80% predicted)
* Subjects are able to give informed consent

Inclusion Criteria-COPD patients (stage II-III according to the GOLD guidelines)

* Current and/or ex-smokers with no less than 10 pack-year smoking history
* aged 40 -75 years
* FEV1 greater than or equal to 30% and less than 80% of predicted (the upper value is a prostbronchodilator value)
* FEV1/FVC < 70%
* Patients with stable COPD
* Inhaled Corticosteroid (ICS) treatment, if exists, must be stopped for 2 weeks prior the study treatment
* Long-acting beta2-agonists and theophylline need to be stopped at least 3 days before run-in , but anti-cholinergics will be allowed throughout the study
* The subjects are able to give informed consent

Exclusion Criteria:

Exclusion Criteria-Healthy non-smokers

* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator
* Upper respiratory infection within the last 4 weeks
* Subjects who have received research medication within the previous one month
* Subjects unable to give informed consent
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.

Exclusion Criteria-COPD patients

* Evidence of asthma
* Bronchodilator reversibility > 12%
* Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator
* Patients who have had oral steroids within 8 weeks prior to the screening visit.
* Patients who are already on ICS and in which it is considered unsafe (as judged by the Investigator) to stop this treatment for the study period.
* Patients who have had an exacerbation which required treatment with oral steroids during the last 2 months prior to the screening visit.
* Upper respiratory infection within the last 4 weeks
* Subjects who have received research medication within the previous one month
* Subjects unable to give informed consent
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patients with significant co-morbidities as judged by the investigator
* Any other respiratory disease, which is considered by the investigator to be clinically significant

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
HDAC and HAT activity ratio

SECONDARY OUTCOMES:
Several inflammation and anti-inflammation markers and lung function will be evaluted as shown below.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Barnes, MA DM DSc FRCP, Principal Investigator — Imperial College London; Kazuhiro Ito, PhD, Principal Investigator — Imperial College London; Ian Adcock, PhD, Principal Investigator — Imperial College London; Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom